CLINICAL TRIAL: NCT04631731
Title: Risk Factors of Immune-ChEckpoint Inhibitors MEdiated Liver, Gastrointestinal, Endocrine and Skin Toxicity
Acronym: ICEMELT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Sydney Local Health District (Other)
Collaborators: University of Western Sydney (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Golo Ahlenstiel, Professor of Medicine, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/PID02542
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer, Nonsmall Cell; Renal Cell Carcinoma; Melanoma; Gastric Cancer; Hepatocellular Carcinoma; Endometrial Cancer; Mesothelioma
Keywords: Immune-checkpoint inhibitors; Immunotherapy; Nivolumab; Iplimumab; Pembrolizumab; Atezolizumab; Durvalumab; CTLA-4; PD-1; PD-L1; Tislelizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Melanoma; Stomach Neoplasms; Carcinoma, Hepatocellular; Endometrial Neoplasms; Mesothelioma; Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Single agent PD-1/L1 inhibitor (Experimental)
  Interventions: Diagnostic Test: Blood screening; Diagnostic Test: Tissue screening
- PD-1/L1 inhibitor + CTLA-4 inhibitor (Experimental)
  Interventions: Diagnostic Test: Blood screening; Diagnostic Test: Tissue screening
- Platinum-based chemotherapy + PD-1/L1 inhibitor (Experimental)
  Interventions: Diagnostic Test: Blood screening; Diagnostic Test: Tissue screening
- PD-1/L1 inhibitor + tyrosine kinase inhibitor (Experimental)
  Interventions: Diagnostic Test: Blood screening; Diagnostic Test: Tissue screening
- PD-1/L1 inhibitor + VEGF inhibitor (Experimental)
  Interventions: Diagnostic Test: Blood screening; Diagnostic Test: Tissue screening

INTERVENTIONS:
Diagnostic Test: Blood screening — Blood will be taken in order to elucidate transcriptomic and proteomic differences (1) pre- and post-ICI treatment commencement; (2) in patients with and without immune-related adverse events.
Diagnostic Test: Tissue screening — Archival tumor tissue (FFPE) will be spatially analysed in order to define tissue heterogeneity in tumor samples regarding cancer immune cell transcriptional profiles and correlate it with the occurrence/development of immune-related adverse events.

SUMMARY:
"Risk factors of Immune-ChEckpoint inhibitor MEdiated Liver, gastrointestinal, endocrine and skin Toxicity" (ICEMELT) study is a prospective multicenter cohort study, enrolling patients who are scheduled to receive (1) single agent PD1/L1 inhibitor; (2) PD1/L1 inhibitor plus CTLA4 inhibitor; (3) platinum-based chemotherapy + PD1/L1 inhibitor; (4) PD1/L1 inhibitor and tyrosine kinase inhibitor and (5) PD1/L1 inhibitor and vascular endothelial growth factor (VEGF) inhibitor.

DETAILED DESCRIPTION:
This project is based on strong multidisciplinary collaboration between oncologists, gastroenterologists/hepatologists, immunologists and basic scientists affiliated with (1) Western Sydney University, (2) University of Sydney, (3) Western Sydney Local Health District (4) New South Wales Health Pathology, (5) Westmead Institute for Medical Research.

Recruitment sites:

* Blacktown Mt Druitt Hospital.
* Westmead Hospital.

Research samples collection, processing and storage:

* Blacktown Clinical School, Western Sydney University.
* Westmead Institute for Medical Research, the University of Sydney.
* New South Wales Health Pathology.

Potential patients will be identified by study investigators at Oncology clinics. After informed consent, clinicopathological data including patients' demographics, past medical history, cancer staging, relevant anticancer treatment, response/progression and survival will be collected longitudinally.

The following specimens will be collected from all participating patients at baseline (pre-treatment stage):

* Peripheral blood (3 x 10mL EDTA tubes)
* FibroScan (CAP score for elucidating pre-existing liver fibrosis)
* Formalin-Fixed Paraffin-Embedded (FFPE) samples (one block) from core biopsies which is a part of routine care for cancer patients.

The following specimens will be collected after IPI + NIVO therapeutic regimen will be commenced (week 6-9 after ICI-therapy commencement):

• Peripheral blood (3 x 10mL EDTA tubes)

Upon development of potential grade ≥2 irAEs, the following samples will be collected:

* Peripheral blood (3 x 10mL EDTA tubes)
* FibroScan (for patients with hepatic irAEs)
* Tissue samples (if biopsies are collected as per standard of care for patients with immune-mediated colitis who will be required to undergo colonoscopy)

Peripheral blood samples from patients will be collected using 10ml EDTA vacutainer tubes (x3) and processed within 12 hours of collection by research staff at each site. Plasma will be used for miRNA assay. PBMCs will be split into 5 cryotubes and used for flow cytometry and single-cell sequencing.

Consent to the study will allow researchers to access the baseline archive diagnostic FFPE tissue samples. With implementing cutting-edge spatial analysis we aim to elucidate the impact of tumour-infiltrating immune microenvironment on clinical outcomes of ICI therapy.

Fresh tissue samples obtained from patients with severe immune-mediated colitis will be processed to obtain total RNA and immune cells for sequencing and mass spectrometry (CyTOF). In addition, tissue samples will be analysed with in situ spatial profiling technologies to map multi-omic data on subcellular level and to determine its association with the clinical outcomes of cancer immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend the requirements and procedures for the study and to provide informed consent before entering the study
* Solid malignant tumour (stage III-IV)
* Treated with ICI-based therapeutic regimens

Exclusion Criteria:

* Inability to give written informed consent
* Patients with a cognitive impairment, an intellectual disability or a mental condition that will interfere with the patient's ability to understand the requirements of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Differentially expressed genes in circulating immune cells between patients with and without irAEs. | Week 0-48
  This objective will be achieved through single-cell sequencing.
Expression of TIM-3, LAG3, VISTA and other inhibitory checkpoint molecules on tumour-infiltrating T cells. | Week 0-48
  In order to ascertain this result, our objective is to utilize spatial transcriptomics and mass spectrometry.

SECONDARY OUTCOMES:
Association of pre-treatment BMI, neutrophil-to-lymphocyte ratio and other clinical parameters with irAEs. | Week 0-48

CONTACTS AND LOCATIONS:
Overall Officials: Golo Ahlenstiel, Professor, Principal Investigator — Western Sydney Local Health District
Locations (2):
- Australia (2):
  - Westmead Hospital, Sydney, New South Wales
  - Blacktown Mt Druitt Hospital, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shek D, Read SA, Akhuba L, Qiao L, Gao B, Nagrial A, Carlino MS, Ahlenstiel G. Non-coding RNA and immune-checkpoint inhibitors: friends or foes? Immunotherapy. 2020 May;12(7):513-529. doi: 10.2217/imt-2019-0204. Epub 2020 May 7. PMID 32378480
- [Background] Shek D, Read SA, Nagrial A, Carlino MS, Gao B, George J, Ahlenstiel G. Immune-Checkpoint Inhibitors for Advanced Hepatocellular Carcinoma: A Synopsis of Response Rates. Oncologist. 2021 Jul;26(7):e1216-e1225. doi: 10.1002/onco.13776. Epub 2021 Apr 21. PMID 33818870
- [Background] Shek D, Akhuba L, Carlino MS, Nagrial A, Moujaber T, Read SA, Gao B, Ahlenstiel G. Immune-Checkpoint Inhibitors for Metastatic Colorectal Cancer: A Systematic Review of Clinical Outcomes. Cancers (Basel). 2021 Aug 27;13(17):4345. doi: 10.3390/cancers13174345. PMID 34503155
- [Result] Shek D, Gloss B, Lai J, Ma L, Zhang HE, Carlino MS, Mahajan H, Nagrial A, Gao B, Read SA, Ahlenstiel G. Identification and Characterisation of Infiltrating Immune Cells in Malignant Pleural Mesothelioma Using Spatial Transcriptomics. Methods Protoc. 2023 Mar 28;6(2):35. doi: 10.3390/mps6020035. PMID 37104017